CLINICAL TRIAL: NCT01399905
Title: A Randomized Controlled Trial of Four Week Outpatient Treatment of Parkinson's Disease Comparing High and Low Dose Carbidopa.
Brief Title: High and Low Dose Carbidopa Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, John G. Nutt, Director, Parkinson Center of Oregon, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00004133; NCT00745277 (obsolete NCT alias)
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Levodopa; Carbidopa; Blood brain barrier
MeSH Terms: conditions — Parkinson Disease | interventions — Carbidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High carbidopa followed by low carbidopa (Experimental): 450 mg of carbidopa per day for four weeks followed by 75 mg of carbidopa per day for four weeks
  Interventions: Drug: carbidopa
- Low carbidopa followed by high carbidopa (Experimental): 75 mg of carbidopa per day for four weeks followed by 450 mg of carbidopa per day
  Interventions: Drug: carbidopa

INTERVENTIONS:
Drug: carbidopa — 75 mg of carbidopa per day versus 450 mg of carbidopa per day

SUMMARY:
Hypothesis: We hypothesize that carbidopa in daily doses of 450mg will enter the central nervous system and partially inhibit AAAD, thereby reducing the decarboxylation of exogenous levodopa to dopamine, and thereby blunt the therapeutic effects of levodopa in PD subjects.

The purpose of this study is to see how low dose vs. high dose of the study drug, carbidopa effect movement in subjects with Parkinson's disease. The low dose of the study drug is 75 mg and the high dose is 450mg.

Subjects will be recruited from the investigators clinic when they are seen for treatment for Parkinson's disease. Subjects will also be recruited through flyers hung at OHSU and at the VA.

Subjects will take part in 2 screening visits one week apart to determine eligibility. Subjects will be randomly chosen to start either high or low dose carbidopa and take it for 4 weeks. Subjects will be called 2, 4, and 6 or 7 days after this visit to ask how they are doing after starting this dose of study drug. We will leave them a message if we cannot reach them. If there are any problems, we will schedule them to come to the clinic within the next 2 days.

Subjects will have an outpatient visit 2 weeks after screening and a hospital admission 2 weeks after that. At the hospital, subjects will stay for 3 days. They will have blood drawn and their Parkinson's disease assessed by a finger tapping exercise, timing their walking, and looking at their uncontrolled movements.

The subject will then receive the opposite dose of carbidopa for 4 weeks. Subjects will be called 2, 4, and 6 or 7 days after this visit to ask how they are doing after starting this dose of study drug. We will leave them a message if we cannot reach them. If there are any problems, we will schedule them to come to the clinic within the next 2 days.

The outpatient visit and hospital admission will repeat again. At the end of the second hospital admission, treatment on the study is over and subjects will go back to their original Parkinson's disease medications. The study will end with a follow up phone call or clinic visit 2 - 4 weeks after the final hospital admission.

Subjects will fill out a daily diary that asks about their movement throughout the day for 3 days before they come to the Oregon Clinical and Translational Research Institute.

Carbidopa is used for the treatment of Parkinson's disease with levodopa. This protocol is using a high dose of 450mg of carbidopa. This study is also using IV levodopa, which is a different route than is normally given.

Finger tapping rates will be compared between high and low dose study drug use to see if one group has slower rates than the other.

DETAILED DESCRIPTION:
A. Specific Aims:

Parkinson's disease is a common neurodegenerative disorder characterized by the progressive motor symptoms of tremor, rigidity, and bradykinesia. The prevalence is estimated at 102-109/100,000 and increases with age. It is the second most common neurodegenerative disorder after Alzheimer's disease, and the annual cost in the US is estimated to be $14.3 billion dollars per year.

In Parkinson's disease (PD) dopamine containing neurons in the substantia nigra are selectively lost, which causes motor dysfunction. Dopamine levels may be increased by giving oral levodopa, which improves motor function in PD. After oral administration, levodopa is taken into the brain and converted into dopamine by aromatic amino acid decarboxylase (AAAD) enzyme in the striatum , resulting in improved dopaminergic neurotransmission. AAAD is found in the peripheral tissues as well as in the brain, and prior to passage into the central nervous system levodopa may be decarboxylated to dopamine in the small bowel and liver. Peripheral metabolism of levodopa to dopamine significantly reduces the amount of levodopa that reaches the brain and therefore dopamine available for neurotransmission. The presence of dopamine in the periphery also produces anorexia and nausea. Carbidopa is an AAAD inhibitor that reduces the conversion of levodopa to dopamine. It is thought to not cross the blood-brain barrier and to affect only peripheral AAAD. This concept is of fundamental importance in the current treatment of PD. Carbidopa potentiates levodopa so that a much lower dose is effective. It also reduces anorexia and nausea, which often occur after giving levodopa alone. For this reason, almost all levodopa is marketed as carbidopa/levodopa tablets. This combination drug has become the standard of care for PD. As the disease progresses, increasingly high amounts of the carbidopa/levodopa combination are given to ensure adequate motor functioning, though the response to treatment becomes much less predictable with frequent fluctuations in motor ability.

Though conventional wisdom and older pharmacological studies suggest carbidopa does not penetrate the blood-brain barrier, recent animal studies contradict this. This is very important because if carbidopa entered the central nervous system in humans it could significantly inhibit levodopa conversion into dopamine, and thus reduce its therapeutic effects. A single large dose of carbidopa given to a normal rat, or a rat chemically lesioned to mimic PD, resulted in carbidopa entrance into the central nervous system, and inhibition of brain AAAD and conversion of levodopa to dopamine (1, 2). It is not known whether prolonged use of high dose carbidopa worsens motor function over time in humans. A small series of patients with PD and motor fluctuations that were switched from carbidopa/levodopa to levodopa alone were reported to have improvement in motor features(3). Carbidopa is typically given in a one to four ratio of carbidopa to levodopa in each pill, and chronic high dosing of caribopa and levodopa is common in PD. If carbidopa penetrates into the central nervous system in humans it could lead to decreased conversion of levodopa to dopamine in the central nervous system, and decrease the therapeutic response to administered levodopa.

We propose a randomized, double blind, controlled trial with crossover to explore two mechanisms by which carbidopa may accumulate in the CNS.

If given in high doses over 4 weeks, carbidopa may slowly accumulate in the central nervous system and impair dopamine synthesis and thereby motor function in PD.

Aim #1: Compare motor response to 2 hour levodopa infusion after 4 weeks of high dose carbidopa and after 4 weeks of low dose carbidopa.

After 4 weeks of high dose carbidopa, subjects may notice more "off" time than after 4 weeks of low dose carbidopa. Changes in response to levodopa can be evaluated by a patient diary and by the need to increase daily levodopa.

Aim 2: Determine the clinical response to oral levodopa at the end of a 4 weeks treatment with high dose carbidopa and with low dose carbidopa measured by an "on/off" diary and with total daily levodopa dose.

An alternate reason for carbidopa to enter the central nervous system (CNS) is through a blood-brain barrier that has become abnormal as a result of age and PD. In this case a single large dose of carbidopa may enter the CNS and reduce the conversion of levodopa to dopamine.

Aim #3: Compare the clinical response to 2 hour levodopa infusion administered with 25mg carbidopa or 150mg carbidopa.

Demonstrating that high doses of carbidopa diminishe the response to levodopa would alter current practice, as clinicians presently are not concerned about the quantity of carbidopa administered to patients with PD. As a result of this study, a significant insight into the management of advanced PD will be gained. The overall goal is to better understand if use of high dose carbidopa may paradoxically complicate treatment. A positive or negative finding will have important therapeutic implications. This study has potential to fundamentally change how we treat PD.

B. Background and Significance:

B. 1 Parkinson's Disease

PD is a common neurodegenerative disorder that results in progressive tremor, rigidity, and bradykinesia. The risk for developing PD increases with age. The prevalence ranges from 102-109/100,000 in Western countries and incidence rate of 1.7 per 1000 person years(4, 5). There is increased direct cost to the individual and a substantial indirect cost to the family(6, 7). The overall estimated cost of PD in the US is $14.3 billion dollars annually(8).

Though PD is associated with a variety of clinical features, patients typically present with motor dysfunction. Motor signs are caused by loss of dopaminergic neurons in the substantia nigra. The mainstay of treatment for motor signs is correction of dopaminergic neurotransmission by oral administration of levodopa, a precursor of dopamine. The risk of death in PD is significantly reduced by the use of levodopa and responsiveness to levodopa treatment is a strong predictor of survival(9, 10).

B. 2. Pharmacology of Levodopa and Carbidopa Levodopa is taken up by the small bowel and heavily metabolized by AAAD located in the intestinal mucosa, and to a lesser degree by the liver. As a result of this first pass peripheral metabolism, the bioavailability of levodopa in the serum after oral administration is approximately 30%(11) and peripheral metabolism of levodopa continues after the first pass metabolism so that only a small amount of levodopa enters the CNS if AAAD is not inhibited. Carbidopa is an AAAD inhibitor and can be given along with levodopa to prevent the peripheral conversion of levodopa to dopamine, and increase the overall bioavailability of levodopa by two to fourfold. Higher doses of carbidopa produce higher plasma levels of levodopa. Carbidopa is also of clinical importance since carbidopa reduces anorexia and nausea related to the effects of dopamine on the area postrema which is effectively outside the blood-brain barrier.

Traditional clinical thinking assumes carbidopa does not penetrate the blood brain barrier, and by this virtue will not interfere with central conversion of levodopa to dopamine (12). The studies supporting this assumption rely on animal models and utilize single doses of carbidopa (13)(14). Clinical dictum indicates a minimum of 75 milligrams of carbidopa be given daily to produce reasonable inhibition of the AAAD. Aside from the primary effect of inhibiting the decarboxylation of levodopa in the periphery and potentiating the effects of levodopa, carbidopa has no demonstrated pharmacological effect. Since carbidopa is not thought to penetrate the blood brain barrier it is considered a peripheral decarboxylase inhibitor.

B. 3. Carbidopa Acts Centrally to Prevent Formation of Dopamine Evidence from laboratory studies has appeared in recent years suggesting carbidopa penetrates the blood brain barrier to a greater extent than realized. One piece of evidence is based on single injection models using microdialysate techniques for drug level measurement in normal rats (1). A single high dose of carbidopa 50mg/kg may inhibit the aromatic amino acid decarboxylase activity in the striatum of normal rats by 75% (2). Benserazide is a peripheral AAAD inhibitor similar to carbidopa. Benserazide administration 50mg/kg prolongs the time to reach peak dopamine level by 60 minutes centrally. Administration of benserazide 10mg/kg and 50mg/kg decreases striatal AAAD activity in normal rats by 28% and 78% respectively, and in rats modeled to mimic PD benserazide 10mg/kg and 50mg/kg decreases striatal AAAD activity 75% and 88%, respectively (15). Even if a small percent of each dose of carbidopa enters the CNS, long-term use could allow carbidopa to accumulate if clearance of carbidopa is not rapid. A small study suggests that motor fluctuations improve in advanced PD when patients receive levodopa without an aromatic amino acid decarboxylase inhibitor (3). It was demonstrated in an earlier study with an experimental formulation of extended release carbidopa/levodopa that some patients had worse motor function with three times the dose of carbidopa/levodopa despite an adequate plasma levodopa level (16). High dose carbidopa is typically used in advanced PD. When high dose carbidopa is given chronically this may create a situation where carbidopa accumulates in the central nervous system and could thereby worsen motor function.

B. 4. Alteration of the Blood Brain Barrier in PD May Be a Mechanism by Which Carbidopa Inhibits Central AAAD Another consideration is that the blood brain barrier is altered in PD and could allow entry of substances previously sequestered to the periphery (17). As PD progresses patients receive larger doses of carbidopa along with levodopa in order to manage motor fluctuations. Chronic levodopa administration often results in dyskinesias in these circumstances. Histochemical evidence from animal models of levodopa induced dyskinesia suggests there is dysfunction of the blood brain barrier. Signs of angiogenesis and serum albumin leakage were two findings supporting vascular alteration in this model (18). Chronic administration of MPTP to primates increases VEGF-expressing neurons and increases the number of blood vessels in the substantia nigra pars comptacta (19). Similarly, in the 6-hydroxydopamine model of PD, primates had patchy loss of blood brain barrier in the same regions associated with angiogenesis (20). In a small autopsy study humans with PD had vascularity present in the substantia nigra pars compacta compared with controls (21). Blood brain barrier alteration could lead to increased penetration of carbidopa from the periphery over time in two different scenarios. Firstly, carbidopa clearing mechanisms and transport pumps may be overwhelmed if small amounts accumulate over time. Secondly, the degree of blood-brain barrier alteration may be so great that even a single large dose of carbidopa may enter the CNS.

Carbidopa penetrates the blood brain barrier to a limited extent after a single injection in normal rats. Since the blood brain barrier could be altered in PD there might be significant inhibition of central AAAD. Either the effect of long-term multiple daily doses of carbidopa or a single large dose of carbidopa could lead to a significant decrease in the amount of available dopamine, thereby worsening the clinical features of PD.

C. Preliminary Studies / Experience of the Investigators:

Our group has extensive experience in randomized controlled clinical trials and proof of principle studies in PD. This includes a large number of levodopa infusion protocols similar to that proposed for the current study. We have recently completed studies examining the dose effect of apomorphine on motor fluctuations (Gunzler in press), clinical testing of concomitantly dosed levodopa and methylphenidate (22), and evolution of response to levodopa over the course of PD (23). We have conducted pilot studies involving both outpatient and Clinical Translational Research Center (CTRC formerly GCRC) admissions for both levodopa and carbidopa (16, 24). Furthermore we have been involved in research on the basic pharmacology and clinical effects of levodopa (25-35).

D. Research Design and Methods

D. 1. Overall Study Design This study will be a randomized, double-blind, \controlled, crossover trial of four week outpatient treatment periods with levodopa and either carbidopa 450mg daily or carbidopa 75mg daily plus placebo (figure 1). Levodopa will be dosed separately in individual capsules at doses and intervals that maximize motor function. Subjects will be selected based on inclusionary and exclusionary criteria and randomized to start in either high dose carbidopa group or low dose carbidopa group. After randomization subjects will be given four weeks of outpatient treatment with levodopa and either high dose carbidopa or low dose carbidopa plus placebo. After this four week treatment phase subjects will be brought into the Clinical Translational Research Center at OHSU (CTRC) for a total of three days. Included in this will be two days measuring objective motor function with levodopa infusion along with a different dose of carbidopa on each of the two days. The evening of admission to the CTRC subjects will turn in ratings of outpatient clinical state collected in a structured diary. After this visit they will crossover and alternately receive either high dose carbidopa or low dose of carbidopa for another four weeks. They will again be brought into the CTRC for a second two day measurement of motor function with levodopa infusion and a different dosing schedule of carbidopa on each of the two days. They will again turn in ratings of outpatient clinical state collected in a structured diary. Both subjects and investigators will remain blinded to the dose of carbidopa for both outpatient phases and one of the two days of each inpatient phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Treatment with carbidopa/levodopa
* Motor fluctuations

Exclusion Criteria:

* Dementia
* Hallucinations
* Age greater than 85

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John G Nutt, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Movement Disorders Clinic at Oregon Health and Science University in Portland, Oregon.
Pre-assignment Details: Of the 17 subjects screened, 14 subjects met enrollment criteria and were randomized into one of the two treatment arms.
Groups:
- Low Carbidopa Followed by High Carbidopa: 75 mg of carbidopa per day for four weeks followed by 450 mg of carbidopa per day for four weeks
Period: Overall Study
Arm/Group | Low Carbidopa Followed by High Carbidopa | High Carbidopa Followed by Low Carbidopa
Started | 7 | 7
Completed | 6 (Subject withdrew from the study before receiving treatment.) | 6 (Subject was treated at least one dose of carbidopa before withdrawing from the study.)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Carbidopa Followed by High Carbidopa | High Carbidopa Followed by Low Carbidopa | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (6) | 65 (5) | 63 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Tapping Speed
Description: Tapping speed is an index of bradykinesia and is used as a response to levodopa infusion.
  Reported as increase over average of three measurements between 8 AM and 9 AM (baseline tapping speed) as (taps/min)*(hours) for tapping scores from beginning of levodopa infusion to 3 hours after conclusion of levodopa infusion.
Time Frame: Performed every 30 minutes from 8 AM to 2 PM
Population: All 12 participants who completed the study were included in the data analysis. Each arm contains data from all 12 participants because this is a cross-over study. All participants participated in both the high-dose and low-dose carbidopa arms.
Measure: Mean (Standard Deviation); unit: (taps/min)*(hours)
Groups:
- Low-dose Carbidopa (75 mg/Day) Day 1: Day 1 of levodopa infusions following 4 weeks of low-dose carbidopa (75 mg/day). Carbidopa 25 mg administered at 8 AM, 10 AM and 12 PM for day 1 infusion.
- Low-dose Carbidopa (75 mg/Day) Day 2: Day 2 of levodopa infusions following 4 weeks of low-dose carbidopa (75 mg/day). Carbidopa 25 mg administered at 8 AM, 10 AM, and 12 PM for day 2 infusion.
- High-dose Carbidopa (450 mg/Day) Day 1: Day 1 of levodopa infusions following 4 weeks of high-dose carbidopa (450 mg/day). Carbidopa 25 mg administered at 8 AM 10 AM and 12 PM for day 1 infusion.
- High-dose Carbidopa (450 mg/Day) Day 2: Day 2 of levodopa infusions following 4 weeks of high-dose carbidopa (450 mg/day). Carbidopa 150 mg administered at 8 AM, 10 AM and 12 PM for day 2 levodopa infusion.
Arm/Group | Low-dose Carbidopa (75 mg/Day) Day 1 | Low-dose Carbidopa (75 mg/Day) Day 2 | High-dose Carbidopa (450 mg/Day) Day 1 | High-dose Carbidopa (450 mg/Day) Day 2
Number analyzed (Participants) | 12 | 12 | 12 | 12
(taps/min)*(hours) | 141 (103) | 141 (131) | 145 (123) | 201 (214)

2. Secondary Outcome: AUC of Levodopa Plasma Concentrations Above Baseline
Description: Baseline value is levodopa concentration at 9 AM. AUC is calculated as levodopa concentrations minus 9 AM value at 30 minute intervals until 2 PM.
Time Frame: Measured every 30 minutes from 9 AM until 2 PM
Population: The levodopa plasma samples of one subject were accidently thawed so samples from 11 participants were used in this data analysis.
Measure: Mean (Standard Deviation); unit: (µg/ml)*(hours)
Groups:
- High-dose Carbidopa (450 mg/Day) Day 1: Day 1 of levodopa infusions following 4 weeks of high-dose carbidopa (450 mg/day). Carbidopa 25 mg administered at 8 AM, 10 AM and 12 PM for day 1 infusion.
- Low-dose Carbidopa (75 mg/Day) Day 2: Day 2 of levodopa infusions following 4 weeks of low-dose carbidopa (75 mg/day). Carbidopa administered at 8 AM, 10 AM and 12 PM for day 2 infusion.
- High-dose Carbidopa (450 mg/Day) Day 2: Day 2 of levodopa infusions following 4 weeks of high-dose carbidopa (450 mg/day). Carbidopa 150 mg administered at 8 AM, 10 AM and 12 PM on day 2.
Arm/Group | Low-dose Carbidopa (75 mg/Day) Day 1 | High-dose Carbidopa (450 mg/Day) Day 1 | Low-dose Carbidopa (75 mg/Day) Day 2 | High-dose Carbidopa (450 mg/Day) Day 2
Number analyzed (Participants) | 11 | 11 | 11 | 11
(µg/ml)*(hours) | 5.38 (1.38) | 5.91 (1.64) | 5.23 (1.23) | 6.13 (1.45)

ADVERSE EVENTS:
Groups:
- Low-dose Carbidopa (75 mg/Day): Due to the cross-over study design all 12 participants who completed the study are included in both the high-dose and low-dose treatment arms.
- High-dose Carbidopa (450 mg/Day): Due to the cross-over study design all 12 participants who completed the study are included in both the high-dose and low-dose treatment arms. In addition, the subject who initiated treatment but did not complete the study is included in this arm for the purpose of reporting adverse events.
Arm/Group | Low-dose Carbidopa (75 mg/Day) | High-dose Carbidopa (450 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 11/12 | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Low-dose Carbidopa (75 mg/Day) (N=12) | High-dose Carbidopa (450 mg/Day) (N=13)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Body aches (General disorders) | 0 (0) | 1 (1)
Difficulty swallowing study drug (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — worsening hypersensitivity pneumonitis
Falls (General disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 3 (3) | 0/12 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Increased dyskinesia (Nervous system disorders) | 1 (1) | 5 (5)
Mania/anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
More off time/tremor (Nervous system disorders) | 10 (10) | 5 (5)
Orthostasis (Cardiac disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice fading (Ear and labyrinth disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small study with limited quantity of patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No